CLINICAL TRIAL: NCT00500409
Title: Safety and Efficacy of OSTEOFORM (rhPTH [1-34]) in Increasing Bone Mineral Density in Osteoporosis. A Randomized Controlled Open-label Multicentre Study in India
Brief Title: Safety and Efficacy of OSTEOFORM (rhPTH [1-34]) in Increasing Bone Mineral Density in Osteoporosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Virchow Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VB006/05
Record Dates: First submitted 2007-07-11; First posted 2007-07-12 (Estimated); Last update posted 2014-12-16 (Estimated); Status verified 2007-07

CONDITIONS: Osteoporosis
Keywords: rhPTH(1-34); Osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — Calcium; Vitamin D

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Drug Group (Experimental): Osteoform
  Interventions: Drug: Osteoform
- Control group (Active Comparator): SHELCAL
  Interventions: Drug: SHELCAL

INTERVENTIONS:
Drug: Osteoform — Administer Osteoform 20 µg daily subcutaneously and 1000 mg calcium and 500 IU vitamin D orally for 180 days
  Arms: Drug Group
Drug: SHELCAL — Administer calcium and vitamin D (1000 mg calcium and 500 IU vitamin D) orally for 180 days
  Other Names: Calcium and vitamin D
  Arms: Control group

SUMMARY:
OSTEOFORM, containing recombinant (rhPTH [1-34]), enhances bone mineral density and reduces risk for vertebral fracture. This study evaluates the safety and efficacy of OSTEOFORM in the treatment of osteoporosis in post-menopausal women.

DETAILED DESCRIPTION:
207 post-menopausal women were enrolled for screening at 6 centres, and supplemented with daily 1000 mg elemental calcium and 500 IU of vitamin D for 45 days. 82 eligible women with osteoporosis were randomly received daily either calcium and vitamin D alone (control group) or Osteoform 20 µg subcutaneously with calcium and vitamin D (drug group) for 12 months. End points such as percentage of increase in bone mineral density and, changes in bone biomarkers (serum osteocalcin, bone specific alkaline phosphatase, and urinary DPD) were evaluated at baseline, and 6 and 12 months after supplementation. Besides, safety parameters and adverse events were monitored through out the study period.

ELIGIBILITY:
Inclusion Criteria:

Postmenopausal women with osteoporosis (Lumbar spine or femoral neck BMD or total hip T-score less than or equal to-2.5)

Exclusion Criteria:

1. Women with vertebral (L1-L4) abnormalities that preclude accurate measurement by DEXA.
2. Women on medications that are known to affect bone for more than 7 days in the past 6 months.
3. Currently taking systemic prednisone, inhaled steroids, anticoagulants, anticonvulsants.
4. History of rhPTH use or known hypersensitivity to study drug.
5. Vitamin D3 deficiency (Vitamin D3 < 20 ng/ml).
6. Abnormal thyroid function.
7. History of kidney disease.
8. Any history of hypercalciuria, hypercalcemia or hyperparathyroidism.
9. History of active or treated tuberculosis or significant liver disease or gastrointestinal disease or cancer.

Ages: 45 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2005-12; Primary Completion 2006-12 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Percentage of change in Bone Mineral Density at lumber spine (L1-L4) in postmenopausal women with osteoporosis at the end of 6 and 12 months. | 6 and 12 months

SECONDARY OUTCOMES:
Percentage of change from baseline in biomarkers of bone formation and bone resorption at the end of 3, 6 and 12 months. | 3, 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Bipin Kumar Sethi, MD, DM, Principal Investigator — CARE Hospitals, Hyderabad, AP, India; Dr. Manoj Chadha, MD, DM, Principal Investigator — P.D. Hinduja Hospital and Medical Research Centre, Mumbai, India; Dr. K.Prasanna Kumar, MD, DM, Principal Investigator — M.S. Ramaiah Medical College, Bangalore, India; Dr. K.D. Modi, MD, DM, Principal Investigator — Medwin Hospital, Hyderabad, AP, India; Dr. Rabinderanath Mehrotra, MD, DM, Principal Investigator — Apollo Hospitals, Hyderabad, AP, India; Dr. Usha Sriram, MD, DM, Principal Investigator — Apollo Hospitals, Chennai, India
Locations (6):
- India (6):
  - Apollo Hospitals, Hyderabaad, Andhra Pradesh
  - CARE Hospitals, Hyderabaad, Andhra Pradesh
  - Medwin Hospital, Hyderabaad, Andhra Pradesh
  - MS Ramaiah Medical College, Bangalore, Karnataka
  - P.D. Hinduja Hospital and Medical Research Center, Mumbai, Maharashtra
  - Apollo Hospitals, Chennai, Tamil Nadu

REFERENCES:
- [Derived] Sethi BK, Chadha M, Modi KD, Kumar KM, Mehrotra R, Sriram U. Efficacy of teriparatide in increasing bone mineral density in postmenopausal women with osteoporosis--an Indian experience. J Assoc Physicians India. 2008 Jun;56:418-24. PMID 18822620